CLINICAL TRIAL: NCT00950131
Title: Testing the Effect of a Warning About New Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: White River Junction Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Attorney General Consumer & Prescriber Education Grant (Other)
Responsible Party: Lisa M. Schwartz, MD, MS, White River Junction VAMC
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 16784
Record Dates: First submitted 2009-07-30; First posted 2009-07-31 (Estimated); Last update posted 2010-04-09 (Estimated); Status verified 2009-07

CONDITIONS: Risk Communication

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Directive new drug warning (Experimental): Survey contains information about when the drug was approved by the FDA (2009)and a directive warning (i.e., stating the issue and why it matters) for new drugs.
  This directive warning mentions that serious drug side effects may emerge only after the drug is already on the market, and the reader should ask their doctor there is an available drug with a longer track record.
  Interventions: Other: Presentation of information about drug approval and level of warning
- Non-directive new drug warning (Experimental): Survey contains information about when the drug was approved by the FDA (2009) and a non-directive warning (i.e., just stating the issue) for new drugs.
  This non-directive warning mentions only that serious drug side effects may emerge only after the drug is already on the market.
  Interventions: Other: Presentation of information about drug approval and level of warning
- No new drug warning (Experimental): Survey contains information about when the drug was approved by the FDA (2009) only.
  Interventions: Other: Presentation of information about drug approval and level of warning

INTERVENTIONS:
Other: Presentation of information about drug approval and level of warning — Presentation of information about date of drug approval with no new drug warning, a non-directive drug box warning or a directive drug box warning

SUMMARY:
The purpose of this study is to test whether a new drug warning decreases enthusiasm for new drugs.

ELIGIBILITY:
Inclusion criteria

* Participants will be randomly selected from a research panel of more than 60,000 U.S. households (Knowledge Networks).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2944 (Actual)
Dates: Start 2009-08; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Hypothetical choice of old (vs. newer) drug | 0 weeks (assessed during intervention)

SECONDARY OUTCOMES:
Comprehension of the drug warning and drug information | 0 weeks (assessed during intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Schwartz, MD, MS, Principal Investigator — White River Junction Veterans Affairs Medical Center; Steven Woloshin, MD, MS, Principal Investigator — White River Junction Veterans Affairs Medical Center

REFERENCES:
- [Derived] Schwartz LM, Woloshin S. Communicating uncertainties about prescription drugs to the public: a national randomized trial. Arch Intern Med. 2011 Sep 12;171(16):1463-8. doi: 10.1001/archinternmed.2011.396. PMID 21911629